CLINICAL TRIAL: NCT02933073
Title: A Phase I Study of Oncoimmunome for the Treatment of Stage III/IV Ovarian Carcinoma
Brief Title: Study of Oncoimmunome for the Treatment of Stage III/IV Ovarian Carcinoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study recruitment is temporary on hold by the sponsor due to patient recruitment challenges and the ongoing review of the investigational adjuvant.
Sponsor: UConn Health (Other)
Responsible Party: Principal Investigator, Susan Tannenbaum, Associate Professor, UConn Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Q16-158-3
Record Dates: First submitted 2016-09-20; First posted 2016-10-14 (Estimated); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- OncoImmunome/Vaccine Phase (Experimental): Women with Stage III/IV Ovarian Cancer who have received the standard of care treatment (surgical debulking and chemotherapy) for their cancer and are now in clinical remission will be given the experimental drug (vaccine) called OncoImmunome, which has been produced specifically for each participant.
  Interventions: Biological: OncoImmunome

INTERVENTIONS:
Biological: OncoImmunome — The OncoImmunome will be a substance composed of a mixture of seven to ten peptides each containing 17-18 amino acids. Given that the vaccine will be tumor-specific based upon mutant peptide sequences identified in each tumor transcriptome, the vaccine for each patient will likely be a unique composition.

SUMMARY:
This is a Phase I trial to test the safety and feasibility of OncoImmunome vaccine in stage III/IV ovarian cancer patients. OncoImmunome is a tumor specific vaccine formulation which is predicted to elicit tumor-protective immune responses. A total of 15 patients will be enrolled from the Principal Investigator (PI) clinical practice. These patients will have just successfully completed standard of care surgical debulking with preservation of fresh tumor, chemotherapy treatment and be in documented clinical remission prior to receiving the vaccine. The patients receive 6-monthly doses of the vaccine and are monitored for up to 5 years post vaccination. This is a personalized vaccine, unique to each patient and is the "first in human" use.

DETAILED DESCRIPTION:
The study will be conducted under an IRB approval, in accordance with FDA regulations and Human Subject Protection regulations. Female patients will undergo standard of care therapy to include exploratory laparotomy and cytoreduction (debulking) surgery followed by chemotherapy. Only patients with histological confirmation of FIGO Stage III/IV epithelial adenocarcinoma of ovarian, tubal or peritoneal origin will be screened and enrolled into the study. At cytoreduction surgery a portion of the surgically resected tumor is preserved for vaccine production. The surgically resected tumor as well as normal cells obtained from peripheral blood shall be used for extraction of RNA and DNA sequencing of the tumor and normal transcriptomes, as well as normal exome sequencing, in the Genomic Core Facility at UConn Health. Patient's blood cells shall also be HLA typed.

When the patient has recovered from surgery, standard of care chemotherapy is given. Following completion of standard chemotherapy (6-8 cycles) and Investigator's confirmation of clinical remission, patients will be consented as subjects for the experimental investigative portion of the study.

The overall purpose of this research study is to produce and test the safety of a new experimental vaccine called OncoImmunome in people with Stage III/IV Ovarian Cancer. An "experimental vaccine" is a vaccine that is being tested and is not approved for sale in the United States by the U.S. Food and Drug Administration (FDA). The study has been divided into two parts: 1)Tumor Tissue and Blood Sample Collection and 2) Vaccine and Follow-up.

Study participants will consent to the following:

1. Tumor Tissue and Blood Sample Collection: The purpose of this part of the study is to collect participants' blood and tumor tissue and test it for genetic mutations. These test results will be used to manufacture a study vaccine that is unique to the participant and to their ovarian cancer.
2. Vaccine and Follow-up: The purpose of this part of the study is to test the safety of the experimental drug (vaccine) called OncoImmunome, which has been produced specifically for each participant.

Subject participation in this research study will last up to 5 years. The vaccine will be produced over a 6 month period, and for six months subjects will receive the study vaccine (1 study vaccine dose per month or 6 study vaccine doses total). However, the researchers will continue to collect all subjects information for up 5 years from the time they provided their tumor sample and blood for the research.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients >18 years of age must have a diagnosis of histologically confirmed Stage III/IV epithelial ovarian/fallopian tube/primary peritoneal adenocarcinoma who have not received any treatment or patients with recurrent Stage III/IV epithelial ovarian/tubal/peritoneal carcinoma with first recurrence ≥12 months after initial therapy and with resectable disease.
2. All patients must have cytoreduction/laparoscopic surgery at UConn Health and their tissue must be stored in the UConn Health Center Research Tissue Registry/Repository (Biorepository) using cryopreservation methods.
3. Patient must have completed standard platinum based adjuvant chemotherapy as per standard-of-care (only applicable for Vaccine Phase).
4. Patients must have a life expectancy of at least 6 months.
5. In the clinical judgment of the investigator, patients must have adequate renal, hepatic, and bone marrow function to complete the study:

   * Hematologic function: Absolute neutrophil count (ANC) must be greater than 1000 per mcl. White blood count equal to or greater than 3000 per mcl, platelet count greater than or equal to 100,000 per mcl.
   * Renal function: Serum creatinine equal to or less than 2.0 mg/dl.
   * Hepatic function: Bilirubin <1.5 x institutional normal.
6. Patients with Patients with ECOG/WHO/Zubrod scale performance status < or = 2.
7. No evidence of active infection.
8. No evidence of active infection requiring systemic therapy. Patients enrolled in the Tissue and Blood Phase may receive IV antibiotics preoperatively, IV in surgery when they have a Hysterectomy and also postoperatively.
9. Patients not participating in another experimental program/therapy at least 4 weeks prior to enrollment.
10. Patients have enrolled and have adequate cancer tissue sample available from this cytoreduction/laparoscopic surgery deposited in the UConn Health Center Research Tissue Registry/Repository (Biorepository) study (Principal Investigator: Mary Melinda Sanders, MD; UConn Health IRB# 08-310-1) for this study.
11. Patients must be English speaking and sign an approved informed consent form (ICF) and HIPAA.

Exclusion Criteria:

1. Patient not enrolled in the UConn Health Center Research Tissue Registry/Repository (Biorepository) study or there is inadequate tissue available for this study.
2. Patients not in clinical remission after standard chemotherapy.
3. Patients with recurrent Stage III/IV epithelial ovarian/tubal/peritoneal carcinoma with first recurrence < 12 months after initial therapy.
4. Patients who have active autoimmune disease.
5. Patients with any medical condition that would interfere with their ability to complete the study.
6. Patients who are receiving any experimental drug therapy within 4 weeks of enrollment.
7. Patients who are taking steroids (excludes topical steroids) within 4 weeks of enrollment.
8. Patients with a prior malignancy within the previous 5 years or a synchronous primary cancer (non-melanoma skin cancer or other In Situ cancers are excluded).
9. Patients unable or unwilling to provide informed consent.
10. Patients whose tumors are not able to be sequenced or from which sufficient suitable neo- epitopes are not able to be identified.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-11; Primary Completion 2022-08 (Actual); Study Completion 2022-08 (Actual)

PRIMARY OUTCOMES:
Monitoring of treatment-related adverse events as assessed by CTCAE v4.0 in subjects immunized with Oncoimmunome | 5 years
  Number of Participants with Oncoimmunome Immunization related Adverse Events (AE) as assessed by CTCAE v. 4.03.

SECONDARY OUTCOMES:
Monitoring of subjects immunized with Oncoimmunome for immune response to components of Oncoimmunome | 5 years
  1) Measurement of CD8 T cell proliferation and T cell phenotype in response to the Oncoimmunome peptides in immunized subjects
Monitoring of subjects immunized with Oncoimmunome for progression-free survival. | 5 years
  Progression-free survival of patients immunized with Oncoimmunome.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Tannenbaum, MD, Principal Investigator — UConn Health
Locations (1):
- UConn Health, Farmington, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No